CLINICAL TRIAL: NCT06361641
Title: Functional and Phenotypic Characterization of Monocytes in Myeloproliferative Syndromes-PHEMOP
Brief Title: Functional and Phenotypic Characterization of Monocytes in Myeloproliferative Syndromes
Acronym: PHEMOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC23_0259; AO2721-44 (Other: ANSM)
Record Dates: First submitted 2024-03-12; First posted 2024-04-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Myeloproliferative Neoplasm; Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phemop Cohort (Experimental)
  Interventions: Diagnostic Test: Monocytes signatures in myeloproliferative neoplasms at diagnosis

INTERVENTIONS:
Diagnostic Test: Monocytes signatures in myeloproliferative neoplasms at diagnosis — The monocytes signatures will be perform from a peripheral blood sample. The signature will be derived from (i) surface marker expression, (ii) cytokines profiles, (iii) genes expression.

SUMMARY:
Prospective study for functional and phenotypic characterization of monocytes in philadelphia-negative myeloproliferative neoplasms

DETAILED DESCRIPTION:
Philadelphia-negative myeloproliferative neoplasms (MPN) are clonal disorders of the hematopoietic stem cell characterized by an excessive production of mature myeloid cells. MPNs are characterized by the presence of somatic gain-of-function mutations present in more than 80% of cases and affecting JAK2, CALR or MPL genes. These mutations lead to a constitutive activation of the JAK-STAT signaling pathway at the origin of cell proliferation.

MPN include polycythemia vera (PV), essential thrombocythemia (ET), prefibrotic primary myelofibrosis (pre-PMF), and primary myelofibrosis (PMF). Despite the classification of MPNs into distinct subtypes based on clinical and pathological features, the precise mechanisms underlying the phenotypic diversity within these disorders remain poorly understood. One aspect that has received limited attention is the role of monocytes and macrophages, key components of the innate immune system, in MPN pathogenesis.

Monocytes, circulating precursors of tissue-resident macrophages, play essential roles in inflammation, immune surveillance, and tissue repair. Upon recruitment to tissues, monocytes differentiate into macrophages with diverse phenotypes and functions influenced by local microenvironmental cues. Macrophages, in turn, exhibit a spectrum of activation states ranging from pro-inflammatory (M1) to anti-inflammatory or pro-repair (M2), with implications for various physiological and pathological processes. Recent studies have implicated monocytes and macrophages in the pathogenesis of MPNs. Circulating monocytes in MPN patients display altered functional characteristics, including dysregulated cytokine production and enhanced fibrotic potential. Additionally, monocytosis, an elevated monocyte count, has been identified as an adverse prognostic factor in MPNs, particularly in PMF.

Based on these observations, investigator propose that monocytes and macrophages contribute to the phenotypic expression of MPNs and that distinct phenotypic and functional signatures of these cells may be associated with different MPN subtypes. By leveraging available techniques for genetic and functional analysis, study team aims to elucidate the role of monocytes and macrophages in MPN pathogenesis and identify potential biomarkers associated with disease phenotype and prognosis. Through comprehensive characterization of these immune cell populations, investigator seek to gain insights into the underlying mechanisms driving the heterogeneity of MPNs and identify novel therapeutic targets for precision medicine approaches.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PV, ET, pre-myelofibrosis or primary myelofibrosis according to WHO 2022 criteria (including BOM for ET, premyelofibrosis and primary myelofibrosis)
* Patient who has not received treatment specific to hemopathy at the time of sampling
* Obtaining the signature of consent to participate in the study
* Patient having consented to be included in the "Malignant Hemopathy" collection of Angers University Hospital and in FIMBANK database

Exclusion Criteria:

* Person not affiliated to a social security scheme or beneficiary of such a scheme
* Patient with another hemopathy or another active cancer at the time of diagnosis
* Minor patient at diagnosis (< 18 years old)
* Patient not capable or without agreement from the guardian or legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2028-10-19 (Estimated)

PRIMARY OUTCOMES:
WHO 2016 criteria for polycythemia vera, prefibrotic myelofibrosis, essential thrombocytosis and overt myelofibrosis diagnosis | Day 0
  Assessment of the monocytic signature against the WHO diagnosis (AUC will be determined)

SECONDARY OUTCOMES:
Identify correlation between the monocytic signature and driver mutations (mutation in JAK2, CALR or MPL gene). | 24 months
  The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis
Identify correlation between the monocytic signature and the grade of fibrosis | 24 months
  The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis The monocytic signature will be compared between the different stages of fibrosis (WHO definition for fibrosis grading)
prognostic value of the monocytic signature using a principal component analysis Response criteria according to Barosi et al., Leukemia, vol. 29,1 (2015): 20-6 | 12, 24 months
  Evaluate the prognostic value of the monocytic signature for treatment response
  The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis Response criteria according to Barosi et al., Leukemia, vol. 29,1 (2015): 20-6 :
  * Complete response: normal blood counts
  * Partial response: platelets between 400 and 600 G/L
  * No response: absence of complete or partial response
Prognostic value of the monocyte signature for disease worsening according to Sureau et al., Blood Cancer Journal, vol. 12,4, 56. 8 Apr. 2022 | 24 months
  Evaluate the prognostic value of the monocyte signature for disease worsening The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis
  Disease worsening criteria according to Sureau et al., Blood Cancer Journal, vol. 12,4, 56. 8 Apr. 2022):
  - Worsening is defined by the presence of at least one of the following criteria: i) leukocytosis >12 G/L or presence of immature granulocytes >2% or erythroblasts >1%; (ii) anemia (hemoglobin <12 g/dL in a woman or <13 g/dL in man) not related to treatment toxicity; (iii) thrombocytopenia (platelet count <150G/L) not related to treatment toxicity; (iv) onset of splenomegaly or progression of pre-existing splenomegaly; (v) thrombocytosis despite cytoreductive therapy
leukemia-free survival | 24 months
  The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis Outcome measure : leukemia-free survival and myelofibrosis-free survival Evaluate the prognostic value of the monocytic signature for hematological progression (acute myeloid leukemia or myelofibrosis)
myelofibrosis-free survival | 24 months
  The monocytic signature will be derived from surface marker expression, cytokines profile and genes expression using a principal component analysis Outcome measure : leukemia-free survival and myelofibrosis-free survival Evaluate the prognostic value of the monocytic signature for hematological progression (acute myeloid leukemia or myelofibrosis)
Monocytes parameters for hematological progression | 24 months
  Evaluate the prosnostic value of monocytes parameters for hematological progression Hematological free survival wil be evaluated by cox models

CONTACTS AND LOCATIONS:
Overall Officials: Agathe GOUBAND, PharmD, Principal Investigator — University Hospital
Locations (3):
- France (3):
  - GOUBAND Agathe, Angers, Maine et Loire
  - BESCOND Charles, Cholet, Maine et Loire
  - TRUCHAN-GRACZYK Malgorzata, Saumur, Maine et Loire

IPD SHARING:
Plan to Share IPD: Undecided